CLINICAL TRIAL: NCT03849742
Title: Ride to Care - A Pilot Study to Investigate the Clinical and Quality of Life Benefit of Eliminating Transportation Barriers for Disadvantaged Cancer Patients Undergoing Ambulatory Palliative Radiotherapy
Brief Title: Ride to Care - Quality of Life With Transportation for RT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 189820; NCI-2019-00448 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-02-12; First posted 2019-02-21 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Locally Advanced Malignant Neoplasm; Metastatic Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Heath services research (Uber rides) (Experimental): Patients receive Uber rides to and from scheduled radiotherapy appointments for up to 6 months.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Supportive Care

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Supportive Care — Receive Uber rides
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive

SUMMARY:
This trial studies how well Uber health intervention works in eliminating transportation barriers for disadvantaged patients with cancer that has spread to nearby tissue, lymph nodes, or other places in the body, undergoing ambulatory palliative radiotherapy. Uber health intervention provides free transportation to disadvantaged patients and may reduce the amount of missed radiotherapy appointments, patient anxiety, and the amount of unplanned emergency department visits, as well as improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test whether eliminating transportation barriers for disadvantaged cancer patients can reduce the 6-month rate of unplanned emergency department (ED) visits.

SECONDARY OBJECTIVES:

I. To test whether eliminating transportation barriers for disadvantaged cancer patients for the duration of a palliative radiotherapy course will improve prescribed treatment completion rates and reduce treatment delays and overall time to treatment completion.

II. To test whether eliminating transportation barriers for disadvantaged cancer patients for the duration of a palliative radiotherapy course will have an impact on physician choice for therapeutic modality, [3-dimensional conformal radiation therapy (3D CRT) versus intensity-modulated radiation therapy (IMRT) versus stereotactic body radiation therapy (SBRT)] and the fractionation schedules to minimize patient inconvenience.

III. To test whether eliminating transportation barriers for disadvantaged cancer patients for the duration of a palliative radiotherapy course can reduce the short-term (6- months) rate of grade >= 3 radiation related adverse events as measured by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.

IV. To test whether eliminating transportation barriers for disadvantaged cancer patients for the duration of a palliative radiotherapy course can improve the patient?s experience, functional outcome, and overall quality of life as measured by the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)30.

V. To test whether eliminating transportation barriers for disadvantaged cancer patients for the duration of a palliative radiotherapy course can reduce re-treatment rates, improve the progression free survival rates, and overall survival.

VI. To determine if living within San Francisco County versus the surrounding counties (Alameda, Contra Costa, Marin, San Mateo) within the San Francisco Bay Area has an impact on outcomes.

OUTLINE:

Patients receive Uber rides to and from scheduled radiotherapy appointments for up to 6 months.

After completion of study, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (and assent when applicable) obtained from patient or patients's legal representative and ability for patient to comply with the requirements of the study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Histologically confirmed locally advanced or metastatic cancer
* Patients who have received prior courses of radiotherapy are eligible
* If patient answers yes to >= 1/4 of the questions below:

  * In the last six months, have you ever delayed seeing a doctor or getting care?
  * Do you anticipate having a hard time coming to University of California, San Francisco (UCSF) for radiation therapy due to transportation challenges?
  * Does lack of money for transportation expenses (parking, taxi, bus) make it difficult for you to get care quickly for medical problems?
  * Does arranging for transportation (driving yourself, getting neighbor or family to drive you) for your cancer treatments make you anxious or worried?"

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Patients who are living at a facility such as a nursing home or skilled nursing facility
* Patients who do not live within a 30-mile radius of one of the radiation oncology sites at University of California San Francisco (UCSF)
* Patients who are currently receiving or expected to be receive UCSF affiliated transportation services prior to enrollment onto the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-02-04 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of unplanned emergency department (ED) visits | Up to 6 months
  For each enrolled patient, any unplanned ED visit over the six months from consultation/enrollment will be documented as an event.
Rate of unplanned hospital admissions | Up to 6 months
  For each enrolled patient, any unplanned hospital admission the six months from consultation/enrollment will be documented as an event.

SECONDARY OUTCOMES:
Change in mean pain score on the European Organization for Research and Treatment of Cancer quality of life questionnaire 30 (EORTC-QLQ-C30) | Up to 3 years
  The Pain score consists of responses to two items with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the two items that make up the pain scale with a resulting total range of 1-4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the pain scale / item represents a high level of symptomatology / problems.
Change in mean overall global health status score on the EORTC-QLQ-C30 | Up to 3 years
  The global health status score consists of responses to two items with responses ranging from 1="very poor" to 4="excellent". The raw score is calculated by estimating the mean of the two items that make up the global health scale with a resulting total range of 1-7. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the global health status represents a higher quality of life.
Change in functional domain scores on the EORTC-QLQ-C30 | Up to 3 years
  The functional domains measure the quality of life in Physical functioning, Role functioning, Emotional functioning, Cognitive functioning, Social functioning. Scores consists of responses to items with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the items that make up each domains with a resulting total range of 1 - 4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the functional domains represents a high level of functioning
Percentage of participants who completed total treatment | Up to 3 years
  Measured by the number of patients who complete treatment in the total sample of participants.
Median days of treatment delays | Up to 3 years
  Will be tabulated. A Mann-Whitney test will be used to compare the two groups.
Number of participants with a reported treatment delay | Up to 3 years
  Will be measured by the ratio of time elapsed to time expected. Patients are assumed to require 2 business days between referral and consult and 3 business days between consult and treatment start. T1/T0, such that time elapsed (T1) = total days between initial referral and treatment completion. Time expected (T0) = 5 + total days of radiation prescribed .
Number of participants with grade >= 3 acute radiation related adverse events | Up to 3 years
  Treatment-related acute adverse events will be classified using the Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5 and tabulated.
Number of participants with grade >= 3 chronic radiation related adverse events | Up to 3 years
  Treatment-related chronic adverse events will be classified using the Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5 and tabulated.
Percentage of participant requiring re-treatment | Up to 3 years
  Defined as the number of participants who needed to undergo re-irradiation due to recurrence or progression at the treatment site in the total sample.
Overall survival (OS) | Up to 3 years
  Participants will be followed from enrollment until end of study or death, whichever occurs first. OS will be assessed using Cox-proportional Hazard models

CONTACTS AND LOCATIONS:
Overall Officials: Steve Braunstein, MD, PhD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No